CLINICAL TRIAL: NCT06491602
Title: A Study of Clinical Characteristics ,Risk Factors and Outcome of Lupus Nephritis Among Children With Systemic Lupus Erthromatousus in Sohag Univeristy Hospital
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Randa Abdelgawad Hussien, Resident-pediatric department-sohag hospital university, Sohag University
Other Study IDs: Soh-Med-24-06-22MS
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: renal biobsy — analsis of renal biobsy and decide grade of renal affection
  Other Names: abdomial us; laboratory investigation for lupus nephritis

SUMMARY:
systemic lupus erthrematosus is an inflamatory and autoimmune condition characterized by multisystem affection and chronic course with unpredictable flares despite potentially afffecting every oragan . kidney involvment are the most common

ELIGIBILITY:
Inclusion Criteria:

- aim to include all children fulfilling diagnostic criteria

Exclusion Criteria:

* children with other rheumatological disorder neonates chidren with other nephrolgy disorder

Ages: 1 Month to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: all children with diagnostic criteria of SLE atteding to pediatric rheumatology and immunology clinic
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2025-06-24 (Estimated); Study Completion 2025-06-24 (Estimated)

PRIMARY OUTCOMES:
remission of LN | 1 year
  acute on top of chronic
progress to CKD | 1 year
  affection of kidney become perment

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tsokos GC. Systemic lupus erythematosus. N Engl J Med. 2011 Dec 1;365(22):2110-21. doi: 10.1056/NEJMra1100359. No abstract available. PMID 22129255
- [Background] Hiraki LT, Feldman CH, Liu J, Alarcon GS, Fischer MA, Winkelmayer WC, Costenbader KH. Prevalence, incidence, and demographics of systemic lupus erythematosus and lupus nephritis from 2000 to 2004 among children in the US Medicaid beneficiary population. Arthritis Rheum. 2012 Aug;64(8):2669-76. doi: 10.1002/art.34472. PMID 22847366
- [Background] Demir S, Gulhan B, Ozen S, Celegen K, Batu ED, Tas N, Orhan D, Bilginer Y, Duzova A, Ozaltin F, Topaloglu R. Long-term renal survival of paediatric patients with lupus nephritis. Nephrol Dial Transplant. 2022 May 25;37(6):1069-1077. doi: 10.1093/ndt/gfab152. PMID 33826705
- [Background] Hiraki LT, Benseler SM, Tyrrell PN, Hebert D, Harvey E, Silverman ED. Clinical and laboratory characteristics and long-term outcome of pediatric systemic lupus erythematosus: a longitudinal study. J Pediatr. 2008 Apr;152(4):550-6. doi: 10.1016/j.jpeds.2007.09.019. Epub 2007 Nov 5. PMID 18346514